CLINICAL TRIAL: NCT02278289
Title: Comparative Effectiveness of Ultrasound and Paraffin Therapy in Patients With Carpal Tunnel Syndrome: A Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BuddhistTCGHTaipei
Record Dates: First submitted 2014-10-13; First posted 2014-10-29 (Estimated); Results first posted 2021-02-24 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2017-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ultrasound therapy group (Active Comparator): Patients in the ultrasound therapy group were treated with US therapy for 5 minutes each session, twice per week for 8 weeks.
  Interventions: Device: ultrasound
- paraffin therapy group (Active Comparator): Patients in the paraffin therapy group were treated with the dip-and-wrap method of paraffin bath therapy in the hospital twice per week for 8 weeks. The temperature of the paraffin bath was maintained at approximately 55°C
  Interventions: Procedure: paraffin therapy

INTERVENTIONS:
Device: ultrasound — Patients in the ultrasound therapy group were treated with US therapy for 5 minutes each session, twice per week for 8 weeks.
  Arms: ultrasound therapy group
Procedure: paraffin therapy — Patients in the paraffin therapy group were treated with the dip-and-wrap method of paraffin bath therapy in the hospital twice per week for 8 weeks. The temperature of the paraffin bath was maintained at approximately 55°C
  Arms: paraffin therapy group

SUMMARY:
The purpose of this study is to compare the efficacy of combining a wrist orthosis with either ultrasound therapy or paraffin bath therapy in treating carpal tunnel syndrome patients.

DETAILED DESCRIPTION:
The purpose of this exploratory study is to compare the combination of a wrist orthosis with either ultrasound therapy or paraffin bath therapy in the treatment of carpal tunnel syndrome patients. We hypothesized that ultrasound therapy might be more effective than paraffin therapy because it provides both thermal and nonthermal effects.

ELIGIBILITY:
Inclusion Criteria:

* patients to have subjective symptoms (such as pain and/or numbness in the median nerve distribution of the digits or nocturnal pain). Furthermore, patients were required to have either a positive Phalen's sign or a positive Tinel's sign along with electrophysiological evidence of carpal tunnel syndrome.

Exclusion Criteria:

* (1) age younger than 18 years old; (2) underlying medical disorders, such as diabetes mellitus, renal failure, autoimmune disease or hypothyroidism; and (3) pregnancy, previous wrist trauma or surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi Shiung Horng, Principal Investigator — Taipei TzuChi hospital

REFERENCES:
- [Derived] Chang YW, Hsieh SF, Horng YS, Chen HL, Lee KC, Horng YS. Comparative effectiveness of ultrasound and paraffin therapy in patients with carpal tunnel syndrome: a randomized trial. BMC Musculoskelet Disord. 2014 Nov 26;15:399. doi: 10.1186/1471-2474-15-399. PMID 25428566

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ultrasound Therapy Group | Paraffin Therapy Group
Started | 30 | 30
Completed | 24 | 23
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound Therapy Group | Paraffin Therapy Group | Total
Number analyzed (Participants) | 24 | 23 | 47
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.8 (11.2) | 51.9 (8.8) | 50.4 (10.1)
Sex/Gender, Customized [Number; unit: participants]
  Female | 22 | 20 | 42
  Male | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Functional Status Scale of the Boston Carpal Tunnel Syndrome Questionnaire
Description: All of the answers were scored from 1 to 5 according to the patient's clinical condition, such that 1 indicated no symptoms, and 5 indicated the most severe symptoms.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ultrasound Therapy Group | Paraffin Therapy Group
Number analyzed (Participants) | 24 | 23
units on a scale | 1.6 (0.7) | 1.8 (0.9)

2. Secondary Outcome: Symptom Severity Scale of the Boston Carpal Tunnel Syndrome Questionnaire
Description: as for outcome 1
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ultrasound Therapy Group | Paraffin Therapy Group
Number analyzed (Participants) | 24 | 23
units on a scale | 2.1 (0.8) | 1.9 (0.7)

3. Secondary Outcome: Pain Scale
Description: The pain VAS is a continuous scale comprised 10 centimeters (100 mm) in length. 0 indicate no pain, 100 indicate maximum pain.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ultrasound Therapy Group | Paraffin Therapy Group
Number analyzed (Participants) | 24 | 23
units on a scale | 54.2 (22.6) | 50.7 (22.7)

4. Secondary Outcome: Difference of Monofilament Sensory Test (Before and After Treatment)
Description: The Semmes-Weinstein monofilament sensory test was measured by applying force-calibrated nylon filament to the fingertips with the wrist in a neutral supine position A weighted score from 1 to 5 was acquired according to each filament's calculated force . We recorded the scores from seven sample areas in each hand and summed the scores to analyze as a continuous variable.Higher score indicate decreased finger tip sensation with increased disesase severity.Total score range:7 -35.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ultrasound Therapy Group | Paraffin Therapy Group
Number analyzed (Participants) | 24 | 23
units on a scale | 1.2 (3.3) | 1.2 (3.5)

5. Secondary Outcome: Difference in Palmar Pinch Power Test (Before and After Treatment)
Description: Palmar pinch strength was measured by pressing the thumb and the index finger tip against a standard dynamometer. This procedure was repeated 3 times measuring in kilograms, and a mean score was obtained. Higher score indicate better pinching strength, which indicate less disease severity. Score range: minimum :0 kilogram
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Ultrasound Therapy Group | Paraffin Therapy Group
Number analyzed (Participants) | 24 | 23
kilograms | 0.5 (1.4) | 0.4 (1.8)

6. Secondary Outcome: Difference in the Distal Sensory Latencies of the Median Nerve (Before and After Treatment)
Description: A standard distance (14 centimeter) was maintained between the stimulator and recording electrodes for the sensory nerve conduction studies. Increased distal latency indicate delay of nerve conduction, which imply poor disease progress.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Ultrasound Therapy Group | Paraffin Therapy Group
Number analyzed (Participants) | 24 | 23
milliseconds | 0.03 (1.1) | -0.2 (0.9)

7. Secondary Outcome: Difference in the Distal Motor Latencies of the Median Nerve (Before and After Treatment)
Description: Median motor nerve conduction and distal motor latency were measured by placing a stimulating electrode at the wrist and a recording electrode on the abductor pollicis brevis muscle 8 centimeter from the stimulus electrode. Increased distal latency indicate delay of nerve conduction, which imply poor disease progress.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Ultrasound Therapy Group | Paraffin Therapy Group
Number analyzed (Participants) | 24 | 23
milliseconds | -0.03 (0.6) | -0.3 (0.6)

ADVERSE EVENTS:
Arm/Group | Ultrasound Therapy Group | Paraffin Therapy Group
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23
Other Adverse Events (participants affected / at risk) | 0/24 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes